CLINICAL TRIAL: NCT02835742
Title: Pulmonary Alveolar Proteinosis GM-CSF Inhalation Efficacy Trial in Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Niigata University Medical & Dental Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAGE
Record Dates: First submitted 2016-07-13; First posted 2016-07-18 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Pulmonary Alveolar Proteinosis, Autoimmune
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis, Acquired | interventions — sargramostim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Group1 (Active Comparator): Treatments for Group 1 include GM-CSF inhalation with 250 mcg/day/body of sargramostim (125 mcg BID on Days 1-7, none on Days 8-14) for twelve 2-week cycles.
  Interventions: Drug: Sargramostim
- Group2 (Placebo Comparator): Treatments for Group 2 include placebo inhalation (Placebo BID on Days 1-7, none on Days 8-14) for twelve 2-week cycles.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sargramostim
  Arms: Group1
Drug: Placebo
  Arms: Group2

SUMMARY:
Objective: Determine the safety and efficacy of GM-CSF inhalation in patients with aPAP.

Study Design: multi-center, randomized, double-blind, placebo- controlled, safety/efficacy study.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 16 years and below 80 years (as of the date of registration).
2. Can provide signed informed consent.
3. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures specified in the protocol (including short-term hospital admission).
4. Autoimmune pulmonary alveolar proteinosis diagnosed by both HR-CT and biopsy and/or BAL as well as GM-CSF antibodies in serum positive.
5. PaO2 < 70 mmHg after 5 minutes spine position at room air, or PaO2 < 75 mmHg after 5 minutes spine position at room air and with symptom(s) including cough, sputum and exertional dyspnea

Exclusion Criteria:

1. Diagnosed as secondary or hereditary pulmonary alveolar proteinosis
2. WBC of 12,000/mm3 or more
3. Fever of 38 degree celsius or more
4. Severe edema
5. History of malignant disease within recent 5 years (not applied to the treated cases of uterine carcinoma in situ and local basal cell carcinoma)
6. Complication of cardiovascular diseases including congestive heart failure, angina pectoris, hemorrhagic tendency, etc with severe condition.
7. Complication of respiratory diseases such as pulmonary infectious disease(incl. pulmonary tuberculosis), bronchial asthma, lung fibrosis ,interstitial pneumonitis, or bronchiectasis, in which the evaluations of safety and efficacy of GM-CSF therapy are considered as difficult.
8. History or complication of infectious diseases which require systemic administration of antibiotics, antifungal or antiviral agents within recent 2 weeks.
9. Treatment with other cytokines
10. Pregnant or possibly pregnant women, lactating women, and women who desire to become pregnant during the study period
11. Patients who have been treated with whole-lung lavage, repeated segmental-lung lavage, or rituximab within 6 months before the start of the study (this criterion does not apply to patients for whom 6 months or more have elapsed after their last lavage or rituximab)
12. Severe liver dysfunction (AST > 100 IU/L and/or ALT > 100 IU/L and/or T-bil >3.0mg/dL)
13. Severe renal dysfunction (Ccr < 30 mL/min, calculated by Cockcroft-Gault (CG) formula)
14. Previous experience of severe and unexplained side-effects during aerosol delivery of any kind of medicinal product
15. Treatment with oral or intravenous administration or inhalation of corticosteroids.
16. Treatment with other inhaled drugs.
17. Previously treated with GM-CSF before the start of the study.
18. Demonstrate hypersensitivity to GM-CSF agent.
19. Other patients judged to be inappropriate for the study by the attending physician (e.g., patients who are unlikely to complete treatment or are uncooperative).

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change value of AaDO2 between baseline and 24 weeks | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Niigata University Med & Dental Hospital, Niigata, Japan

REFERENCES:
- [Derived] Tazawa R, Ueda T, Abe M, Tatsumi K, Eda R, Kondoh S, Morimoto K, Tanaka T, Yamaguchi E, Takahashi A, Oda M, Ishii H, Izumi S, Sugiyama H, Nakagawa A, Tomii K, Suzuki M, Konno S, Ohkouchi S, Tode N, Handa T, Hirai T, Inoue Y, Arai T, Asakawa K, Sakagami T, Hashimoto A, Tanaka T, Takada T, Mikami A, Kitamura N, Nakata K. Inhaled GM-CSF for Pulmonary Alveolar Proteinosis. N Engl J Med. 2019 Sep 5;381(10):923-932. doi: 10.1056/NEJMoa1816216. PMID 31483963